CLINICAL TRIAL: NCT02556827
Title: Investigation of Relation Between Demodex Density With Immune Response and Oxidative Stress in Rosacea Patients
Brief Title: Demodex Density, Immune Response and Oxidative Stress in Rosacea Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Training and Research Hospital (Other Government)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Tuğba Falay, Resident Doctor, Istanbul Training and Research Hospital
Other Study IDs: 71306642-050.01.04
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Rosacea
Keywords: demodex; oxidative stress; reflectance confocal microscopy
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- H, Rosacea patients: Rosacea patients who were between the ages of 18-70, having no systemic illness and who were not smoking.
  Obtaining a blood sample; TOC, TAC, OSI, PON-1, ARES, MPO, TNF-α, IL-1β, MMP-1 and MMP-9 levels in venous blood were measured Reflectance confocal microscopy; 1mm2-sized 10 images were taken from right cheek and forehead; the number of demodex, follicle, the number of mite per follicle, the number of infested follicle and the number of mite per infested follicle were calculated with RCM. And photoaging severity were also assessed by using RCM. Sebum rate at forehead and right cheek were evaluated with sebumeter. Dermoscopic photoaging scale were assessed by using video dermoscopy.
  Interventions: Other: Obtaining a blood sample; Device: Reflectance confocal microscopy; Device: Sebumeter; Device: Video dermoscopy
- K, Healthy volunteers: Healthy volunteers who were compatible in terms of age, sex and skin phenotype, having no systemic illness and who were not smoking.
  Obtaining a blood sample; TOC, TAC, OSI, PON-1, ARES, MPO, TNF-α, IL-1β, MMP-1 and MMP-9 levels in venous blood were measured Reflectance confocal microscopy; 1mm2-sized 10 images were taken from right cheek and forehead; the number of demodex, follicle, the number of mite per follicle, the number of infested follicle and the number of mite per infested follicle were calculated with RCM. And photoaging severity were also assessed by using RCM. Sebum rate at forehead and right cheek were evaluated with sebumeter. Dermoscopic photoaging scale were assessed by using video dermoscopy.
  Interventions: Other: Obtaining a blood sample; Device: Reflectance confocal microscopy; Device: Sebumeter; Device: Video dermoscopy

INTERVENTIONS:
Other: Obtaining a blood sample — Total oxidant capacity (TOC), total antioxidant capacity (TAC), oxidative stress index (OSI), paraoxonase-1 (PON-1), aryl esterase (ARES), myeloperoxidase (MPO), tumor necrosis factor-alpha (TNF-α), interleukin-1beta (IL-1β), matrix metalloproteinase-1 (MMP-1) and matrix metalloproteinase-9 (MMP-9) levels in venous blood were measured.
Device: Reflectance confocal microscopy — 1mm2-sized 10 images were taken from right cheek and forehead; the number of demodex, follicle, the number of mite per follicle, the number of infested follicle and the number of mite per infested follicle were calculated with RCM. And photoaging severity were also assessed by using RCM.
Device: Sebumeter — Sebum rate at forehead and right cheek were evaluated with sebumeter
Device: Video dermoscopy — Dermoscopic photoaging scale were assessed by using video dermoscopy.

SUMMARY:
Aim of study is to determine reactive oxygen products and antioxidant capacity with rosacea patients; to measure metalloproteinase level and inflammatory markers of immune response and investigate their corelation with demodex infestation and also investigate the role of photoaging and sebum secretion in rosacea.

DETAILED DESCRIPTION:
Rosacea is a common and chronic inflammatory disease characterized by facial erythema, papule, pustule and telangiectasia. Ultraviolet, Demodex mite, oxidative stress and antioxidant system disorders are emphasized in increased inflammation seen in rosacea.

The aim of our study was to evaluate the status of oxidative stress, matrix metalloproteinase (MMP) and inflammatory markers in systemic circulation, their relationship with demodex density and investigate the role of photoaging and sebum secretion in rosacea.

Forty patients with rosacea and age, gender and skin phenotype matched 40 healthy volunteers were enrolled in the study. Reflectance confocal microscopy (RCM) was used to calculate facial demodex density. The number of demodex, follicle, the number of mite per follicle, the number of infested follicle and the number of mite per infested follicle were calculated with RCM.

Photoaging severity and facial sebum levels were also assessed. Total oxidant capacity (TOC), total antioxidant capacity (TAC), oxidative stress index (OSI), paraoxonase-1 (PON-1), aryl esterase (ARES), myeloperoxidase (MPO), tumor necrosis factor-alpha (TNF-α), interleukin-1beta (IL-1β), matrix metalloproteinase-1 (MMP-1) and matrix metalloproteinase-9 (MMP-9) levels in venous blood were measured.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-70
* No systemic illness
* No other inflammatory dermatoses except for rosacea
* No smoking
* Not using any topical, systemic treatment and sunblock at least a month for rosacea or other condition

Exclusion Criteria:

* Systemic illness
* Other inflammatory dermatoses except for rosacea
* Smoking
* Using any topical, systemic treatment and sunblock for rosacea or other condition
* Type 4 rosacea patient (only ocular involvement)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Rosacea patients who are between the ages of 18-70, who having no systemic illness and who were not smoking and who were not using any topical and systemic treatment for a month attended to the study. As a control group it was planned that healthy volunteers who were compatible in terms of age, sex and skin phenotype, who were not smoking, with no systemic illness to be taken.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Severity of rosacea | Rosacea patients who refer to criteria will be evaluated throughout 4 months.

SECONDARY OUTCOMES:
The number of demodex of right cheek and forehead | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.
The number of follicle of right cheek and forehead | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.
The number of mite per follicle of right cheek and forehead | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.
The number of infested follicle of right cheek and forehead | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.
The number of mite per infested follicle of right cheek and forehead | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.
Total oxidant capacity (TOC) | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.
Total antioxidant capacity (TAC) | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.
Oxidative stress index (OSI) | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.
Paraoxonase-1 (PON-1) | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.
Aryl esterase (ARES) | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.
Myeloperoxidase (MPO) | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.
Tumor necrosis factor-alpha (TNF-α) | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.
Interleukin-1beta (IL-1β) | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.
Matrix metalloproteinase-1 (MMP-1) | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.
Matrix metalloproteinase-1 (MMP-9) | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.

OTHER OUTCOMES:
Sebum levels of right cheek and forehead | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.
Photoaging severity of face by using RCM and dermoscopy | Rosacea patients and healthy volunteers who refer to criteria will be evaluated throughout 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Falay, Principal Investigator — Istanbul Training and Research Hospital; Vefa Aslı Erdemir, Study Director — Istanbul Training and Research Hospital; Mehmet Salih Gürel, Study Director — Istanbul Training and Research Hospital; Abdurrahim Kocyigit, Study Director — Bezmialem Vakif University; Duygu Erdil, Study Chair — Istanbul Training and Research Hospital; Eray Metin Güler, Study Chair — Bezmialem Vakif University
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Org. Abd. Nafiz Gürman, Turkey (Türkiye)